CLINICAL TRIAL: NCT05347693
Title: An Open-Label, Randomised, Phase 4 Study of Continuing Sodium Zirconium Cyclosilicate (SZC) After Discharge in Participants With Chronic Kidney Disease Treated for Hyperkalaemia
Brief Title: Continuing Sodium Zirconium Cyclosilicate (SZC) After Discharge Study
Acronym: CONTINUITY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9480C00023; 2021-003527-14 (EudraCT Number)
Record Dates: First submitted 2022-02-23; First posted 2022-04-26 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hyperkalaemia; Chronic Kidney Disease
Keywords: sodium zirconium cyclosilicate; Hyperkalaemia after discharge at the hospital
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: This is a Phase 4, randomised, controlled, open-label, parallel-group, multicentre study in participants with CKD treated for HK whilst in hospital.
  * During the in-hospital phase, participants will be treated with SZC as per local label
  * At discharge, NK participants who have been treated with SZC for between 1 and 21 days whilst in hospital and are started on SZC maintenance dose will be randomised in a 1:1 ratio to one of the following arms:
    * Arm A: Participants discharged with SZC, as per local label, to manage HK until the end of the outpatient phase
    * Arm B: Participants discharged with SoC, as per local practice, to manage HK until the end of study. Note: Participants intended to be discharged with a K+ binder (as per the site routine medical practice) will not be randomised and will be discontinued from the study.
  * The total duration of the study for each participant will be up to approximately 6 months.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sodium Zirconium Cyclosilicate (SZC) (Experimental): Participants discharged with SZC, as per local label, to manage HK until the end of the outpatient phase
  Interventions: Drug: Sodium Zirconium Cyclosilicate (SZC)
- Local standard of care (SoC) (Active Comparator): Participants discharged with SoC, as per local practice, to manage HK until the end of study.
  Interventions: Drug: Local standard of care

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (SZC) — White to grey crystalline powder for oral suspension in 5 g sachets. Each sachet will be labeled in accordance with Good Manufacturing Practice Annex 13 and per country regulatory requirement.
  Label text will be translated into local language.
  Other Names: Lokelma
  Arms: Sodium Zirconium Cyclosilicate (SZC)
Drug: Local standard of care — Local SoC in the country to be used as per local label
  Other Names: SoC
  Arms: Local standard of care (SoC)

SUMMARY:
This is an open-label, randomised study in participants with chronic kidney disease (CKD) treated for hyperkalaemia (HK) whilst in hospital. The study will compare SZC to standard of care (SoC) with the goal of determining:

* If continued use of SZC maintains normokalaemia (NK) better than SoC after participant discharge from the hospital.
* If continued use of SZC after discharge will reduce HK related healthcare resource utilisation compared to SoC.

DETAILED DESCRIPTION:
This is a Phase 4, randomised, controlled, open-label, parallel-group, multicentre study in participants with CKD treated for HK whilst in hospital.

* Participants from 30 to 50 sites in 4 to 7 countries will be screened for enrolment. In total, up to a maximum of 163 participants will be enrolled, resulting in approximately 130 participants discharged and randomised and 104 evaluable participants (52 per arm).
* The study plans to enrol approximately equal numbers of participants with mild HK (K+ between > 5.0 and ≤ 5.5 mmol/L) and with moderate/severe HK (K+ between > 5.5 and ≤ 6.5 mmol/L), with a minimum of 30% of the enrolled participants in either group.
* During the in-hospital phase, participants will be treated with SZC as per local label, starting at baseline and based on local K+ measurement obtained within 24 hours of treatment initiation:).

  * Participants with HK (K+ between > 5.0 and ≤ 6.5 mmol/L):

    1. stop current K-binder if any
    2. start SZC correction dose (note: participants currently on SZC should continue SZC correction dose, up to 72 hours).
  * Participants currently receiving any treatment for the current episode of HK and are already NK at baseline (K+ ≤ 5.0 mmol/L): 1) stop any current K-binder, 2) start SZC maintenance dose (note: participants currently on SZC maintenance dose should continue SZC maintenance dose).
  * All treatment decisions, including modification of the ongoing therapy for HK must be based on the investigator's medical judgement of the participant's best interest.
* At discharge, NK participants who have been treated with SZC for between 1 and 21 days whilst in hospital and are started on SZC maintenance dose will be randomised in a 1:1 ratio to one of the following arms:

  * Arm A: Participants discharged with SZC, as per local label, to manage HK until the end of the outpatient phase
  * Arm B: Participants discharged with SoC, as per local practice, to manage HK until the end of study. Note: Participants intended to be discharged with a K+ binder (as per the site routine medical practice) will not be randomised and will be discontinued from the study. Still, participants randomised into Arm B may have a K-binder prescribed at Day 7 post-discharge, (or after Day 7 post-discharge), to treat confirmed HK or in case there is an increase in K+ level since discharge that, in the investigator's opinion, requires therapy.
* The total duration of the study for each participant will be up to approximately 6 months.
* Study visit schedule is as follows:

In-hospital phase: - The screening visit will occur while the participant is at the hospital (up to 21 days before discharge; medical monitor's approval may be sought for allowing longer duration hospital stays for specific participants) in order to check eligibility criteria

* Inpatient phase: o The baseline visit (can occur the same day as the screening visit) where treatment with SZC will be initiated

  o The discharge visit, 1 to 20 days after baseline; medical monitor's approval may be sought for allowing longer duration hospital stays for specific participants). Randomisation will occur at day of discharge.
* Outpatient phase: - Visits will occur at 7, 30, 60, 90, 120, 150, and 180 (EOT, End of Trial) days after randomisation. Only visits at 7, 90 and 180 days after randomisation will be on-site visits, the remaining being telephone visits. If dose titration occurs at any time during the outpatient phase, unscheduled dispensation visits will be performed.

Follow-up phase: - A follow-up on-site visit (end of study visit) will occur approximately 7 days after EOT. • Data will be collected at on-site visits, via telephone visits and medical chart reviews.

• An adjudication committee will be involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older, at the time of signing the informed consent
* Admitted to hospital (inpatient care; directly or from ED)
* With:

  1. Diagnosed CKD (any stage) or
  2. eGFR < 90 ml/min/1.73 m2 at, or within 3 months of, study screening, based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (Levey et al, 2009).

Note: Race/ethnicity should not be included in CKD-EPI equation calculation.

* Local laboratory K+ measurement within 24 hours of baseline visit (visit 2), where result is either:
* Hyperkalaemic as defined by site's local practice and K+ ≤ 6.5 mmol/L.
* Or, normokalaemic: K+ between ≥ 3.5 and ≤ 5.0 mmol/L, where patient started and is receiving treatment for this episode of HK
* Male or female
* Capable and willing of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Hospitalisation for an acute cardiovascular event within 12 weeks prior to screening
* Unable to take oral SZC drug mix
* With a life expectancy of less than 6 months
* Any medical condition that, in the opinion of the investigator makes the participant not suitable for inclusion
* QT interval corrected by the Fridericia method (QTcF) > 550 msec
* History of QT prolongation associated with other medications that required discontinuation of that medication
* Congenital long QT syndrome
* Clinically significant arrythmias as judged by the investigator
* Ongoing treatment with SZC or patiromer before current ED visit/hospital admission (ongoing treatment with other K-binders before current ED visit/hospital admission is allowed).

Note: Initiation of any SZC or patiromer during the current ED visit/hospitalisation preceding enrolment is allowed.

* Chronic haemodialysis or peritoneal dialysis or the recipient of or scheduled date for a kidney transplant. Note: Emergency/unscheduled haemodialysis to treat HK during the current ED visit/hospitalisation preceding enrolment is allowed.
* Participation in another clinical study with an investigational medicinal product (IMP) administered during the month before screening.
* Known hypersensitivity to SZC or any of the excipients of the product
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements
* Previous randomisation in the present study
* For women only: Women of child-bearing potential (WOCBP; ie, those who are not chemically or surgically sterilised or who are not post-menopausal) who are not willing to use one of the methods of contraception described hereafter, or who are not stable on the contraception method for the last one month, from the time of signing the informed consent throughout the study and 7 days after the last dose: (a) Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal (b) Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable (c) Intrauterine device (d) Intrauterine hormone-releasing system (e) Bilateral tubal occlusion (f) Vasectomised partner (vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP participant and that the vasectomised partner has received medical assessment of the surgical success (g) Sexual abstinence: it is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.
* For WOCBP only: Women who have a positive pregnancy test at screening OR women who are breastfeeding.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- Belgium (2):
  - Research Site, Bonheiden
  - Research Site, Leuven
- France (4):
  - Research Site, Annonay
  - Research Site, Ars-Laquenexy
  - Research Site, Nice
  - Research Site, Saint-Priest-en-Jarez
- Italy (4):
  - Research Site, Bari
  - Research Site, Foggia
  - Research Site, Parma
  - Research Site, Pavia
- Research Site, Eindhoven, Netherlands
- Spain (12):
  - Research Site, Algeciras
  - Research Site, Almería
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Getafe
  - Research Site, Madrid
  - Research Site, Salamanca
  - Research Site, San Sebastián de los Reyes
  - Research Site, Seville
  - Research Site, Talavera de la Reina
  - Research Site, Zamora
- United Kingdom (4):
  - Research Site, Doncaster
  - Research Site, Hull
  - Research Site, Salford
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Burton JO, Allum AM, Amin A, Linde C, Lesen E, Mellstrom C, Eudicone JM, Sood MM. Rationale and design of CONTINUITY: a Phase 4 randomized controlled trial of continued post-discharge sodium zirconium cyclosilicate treatment versus standard of care for hyperkalemia in chronic kidney disease. Clin Kidney J. 2023 Mar 23;16(7):1160-1169. doi: 10.1093/ckj/sfad053. eCollection 2023 Jul. PMID 37398685
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00023&attachmentIdentifier=85f086a3-3ed8-47fb-8754-eb08ea667f44&fileName=D9480C00023_CSP_redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00023&attachmentIdentifier=8247aa0a-afb5-4609-9281-450c5156d810&fileName=D9480C00023_SAP_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00023&attachmentIdentifier=19a15e12-c692-4461-8a06-f91f9523371e&fileName=D9480C00023_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 186 participants were screened from 28 study sites across 6 countries.
Pre-assignment Details: This study consisted of 2 phases: an inpatient period and an outpatient period.
  Of the 186 participants enrolled in the inpatient period, 137 participants were randomized into the outpatient period (68 to Arm A and 69 to Arm B). The remaining 49 participants were not randomized due to reasons such as withdrawal of consent, failure to meet inclusion/exclusion criteria, screening failure, death, or other reasons (eg, mistaken study termination or discharged without notifying investigators).
Groups:
- Inpatient Period: Participants were treated with SZC as per local label (correction and/or maintenance treatment), starting at baseline and based on local potassium (K+) measurement obtained within 24 hours of treatment initiation.
- Outpatient Period - Arm A: SZC: Participants discharged with SZC, as per local label, to manage hyperkalaemia (HK) until 7 days before the end of the study.
- Outpatient Period - Arm B: Standard of Care (SoC): SZC was withdrawn and participants discharged with SoC, as per local practice, to manage HK until the end of study.
Period: Inpatient Period
Arm/Group | Inpatient Period | Outpatient Period - Arm A: SZC | Outpatient Period - Arm B: Standard of Care (SoC)
Started | 186 | 0 | 0
Completed | 137 | 0 | 0
Not Completed | 49 | 0 | 0
Not completed — Participant was discharged from the hospital but did not inform the site | 1 | 0 | 0
Not completed — Withdrawal of consent | 10 | 0 | 0
Not completed — Failure to meet inclusion/exclusion criteria | 19 | 0 | 0
Not completed — Screening Failure | 8 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Physician Decision | 5 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawn from study due to a mistaken request for study termination | 1 | 0 | 0
Period: Outpatient Period
Arm/Group | Inpatient Period | Outpatient Period - Arm A: SZC | Outpatient Period - Arm B: Standard of Care (SoC)
Started | 0 | 68 | 69
Completed | 0 | 42 | 56
Not Completed | 0 | 26 | 13
Not completed — Adverse Event | 0 | 9 | 0
Not completed — Death | 0 | 6 | 2
Not completed — Development of study-specific withdrawal criteria: Severe HK | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Participant's study compliance was impossible to monitor and they had a complex private situation. | 0 | 1 | 0
Not completed — Scheduled hemodialysis | 0 | 1 | 0
Not completed — Severe HK | 0 | 0 | 1
Not completed — Started dialysis on 16 Feb 2023 | 0 | 1 | 0
Not completed — Start of dialysis | 0 | 0 | 1
Not completed — The participant entered hemodialysis | 0 | 0 | 1
Not completed — The participant moved to another city and could not attend the study visits | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 8 | 5

BASELINE CHARACTERISTICS:
Population: Safety Set Randomized. Of the 137 participants randomised into the 2 arms (68 participants in Arm A: SZC and 69 participants in Arm B: SoC), there was one participant in Arm B: SoC who did not receive treatment during the outpatient period and was excluded from the safety analysis.
Groups:
- Outpatient Period - Arm A: SZC: Participants discharged with SZC, as per local label, to manage HK until 7 days before the end of the study.
- Outpatient Period - Arm B: SoC: SZC was withdrawn and participants discharged with SoC, as per local practice, to manage HK until the end of study.
- Total: Total of all reporting groups
Arm/Group | Outpatient Period - Arm A: SZC | Outpatient Period - Arm B: SoC | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Screening
  Years | 72.8 (10.25) | 72.1 (10.99) | 72.5 (10.59)
Age, Customized [Number; unit: Participants] — Age at Screening
  Participants
    18-64 years | 14 | 13 | 27
    65-84 years | 45 | 47 | 92
    >=85 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 43 | 52 | 95
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 21 | 10 | 31
  Not Hispanic or Latino | 43 | 56 | 99
  Not Reported | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 64 | 64 | 128
  Black or African American | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  American Indian or Alaskan Native | 0 | 0 | 0
  Other | 0 | 0 | 0
  Multiple | 0 | 0 | 0
  Not Reported | 4 | 3 | 7
Country [Number; unit: Participants]
  Belgium | 0 | 2 | 2
  Spain | 57 | 59 | 116
  France | 4 | 2 | 6
  United Kingdom | 0 | 2 | 2
  Italy | 6 | 3 | 9
  Netherlands | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Occurrence (Yes/No) of NK (K+ Between 3.5 and 5.0 mmol/L, Inclusive) at 180 Days Post-discharge
Description: A response was defined as a participant having serum K+ within 3.5 and 5.0 mmol/L at 180 days post-discharge.
  No response was defined as a participant who: 1) used rescue therapy for hyperkalaemia (HK) during the outpatient period; 1) died prior to 180 days post-discharge; 3) were missing an assessment at visit 10; 4) were lost to follow-up prior to 180 days post-discharge; 5) down-titrated (or discontinued) RAASi.
  The number of participants who had a response/no response is presented.
Time Frame: At 180 days post-discharge (Visit 10)
Population: Full Analysis Set (FAS). The FAS included all randomised participants.
Measure: Number; unit: Number of participants
Groups:
- Arm A: SZC: Participants discharged with SZC, as per local label, to manage HK until 7 days before the end of the study.
- Arm B: SoC: SZC was withdrawn and participants discharged with SoC, as per local practice, to manage HK until the end of study.
Arm/Group | Arm A: SZC | Arm B: SoC
Number analyzed (Participants) | 68 | 69
Number of participants
  Response | 21 | 25
  No response | 47 | 44
Statistical Analysis 1: Comparison: Arm A: SZC vs Arm B: SoC; Test type: Equivalence — Prespecified estimates for sample size calculation * Equivalence margin: 0.29 * Sample size estimate parameters: * Two-group χ² test * Significance level (α): 5% (two-sided) * Power: 80% * Assumed proportions with NK (K+ between 3.5 and 5.0 mmol/L, inclusive) at 180 days post-discharge: * Arm A: 0.88 * Arm B: 0.59 Note: Assumed proportions for statistical planning; not actual results; p = 0.558, Regression, Logistic; Model included response as the dependent variable, and randomised treatment and participant recruitment country as independent factors; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.39 to 1.66] — OR >1 indicated increased odds of K+ between 3.5 and 5.0 mmol/L on SZC compared to SoC

2. Secondary Outcome: Time to First Occurrence of Any Component of All-cause Hospital Admissions or ED Visits With HK as a Contributing Factor, or All-cause Death, or Use of Rescue Therapy for HK at Any Time Post-discharge up to 180 Days
Description: The time to first occurrence of all-cause hospital admission, emergency department (ED) visits with HK as a contributing factor, all-cause death or use of rescue therapy for HK was calculated as date of first occurrence of (all-cause hospital admission, ED visits with HK as a contributing factor, all-cause death, use of rescue therapy for HK, date of loss to follow-up) - date of randomization + 1.
  The median time to event (days) is presented.
Time Frame: At any time post-discharge (from Visits 4 to 10), up to 180 days
Population: FAS. The FAS included all randomised participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A: SZC | Arm B: SoC
Number analyzed (Participants) | 68 | 69
Days | 136 [60.00 to NA] — Although over 50% of participants experienced an event, there were proportionally too few events to estimate an upper confidence interval for the median. | NA [63.00 to NA] — Fewer than 50% of participants experienced an event and no median time and upper confidence interval could be calculated.
Statistical Analysis 1: Comparison: Arm A: SZC vs Arm B: SoC; Test type: Equivalence — Prespecified estimates for sample size calculation * Equivalence margin: 0.262 * Sample size estimate parameters: * Log-Rank Test for Equality of Survival Curves * α: 5% * Power: 80% * HR (SZC/SoC): 0.329 * Assumed proportions without the main secondary composite outcome (event-free) at 180 days post-discharge * Arm A: 83% (17% with the outcome/event of interest) * Arm B: 56.8% (43.2% with the outcome/event of interest) Note: Assumed proportions for statistical planning; not actual results; p = 0.743, Regression, Cox; Randomised treatment group and participant recruitment country were used as the independent variables. SoC group used as reference level in Cox model; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.56 to 1.51] — An HR <1 favoured SZC to be associated with a longer time to first component of composite endpoint than SoC

3. Secondary Outcome: Time to First Occurrence of Any Component of All-cause Hospital Admission or ED Visit With HK as a Contributing Factor at Any Time Post-discharge up to 180 Days
Description: The time to first occurrence of any component of all-cause hospital admission or ED visit with HK as a contributing factor at any time post-discharge up to 180 days was calculated as the earliest date of (all-cause hospital admission, ED visits with HK as a contributing factor, all-cause death, use of rescue therapy for HK, date of loss to follow-up, date of 180 days post-discharge) - date of randomization + 1.
  The median time to event (days) is presented.
Time Frame: At any time post-discharge (from Visits 4 to 10), up to 180 days
Population: FAS. The FAS included all randomised participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A: SZC | Arm B: SoC
Number analyzed (Participants) | 68 | 69
Days | NA [116.00 to NA] — Fewer than 50% of participants experienced an event and no median time and upper confidence interval could be calculated. | NA [123.00 to NA] — Fewer than 50% of participants experienced an event and no median time and upper confidence interval could be calculated.
Statistical Analysis 1: Comparison: Arm A: SZC vs Arm B: SoC; Test type: Equivalence — This outcome is unpowered; p = 0.951, Regression, Cox; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.58 to 1.79] — An HR <1 favoured SZC to be associated with a longer time to first component of composite endpoint than SoC

4. Secondary Outcome: Number of All-cause Events (Hospital Admissions or ED Visits) With HK as a Contributing Factor at Any Time Post-discharge up to 180 Days
Description: The number of all-cause events (hospital admissions or ED visits) with HK as a contributing factor at any time post-discharge up to 180 days is presented.
  Participants who discontinued treatment, used rescue therapy for HK, experienced all-cause death or loss to follow-up prior to 180 days post-discharge or who down-titrated (including discontinued) RAASi were to have all available hospital admission data used irrespective of the intercurrent event (treatment policy strategy).
Time Frame: At any time post-discharge (from Visits 4 to 10), up to 180 days
Population: FAS. The FAS included all randomised participants.
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Arm A: SZC | Arm B: SoC
Number analyzed (Participants) | 68 | 69
Events | 0.7 (0.92) | 0.6 (0.83)
Statistical Analysis 1: Comparison: Arm A: SZC vs Arm B: SoC; Test type: Equivalence — This outcome is unpowered; p = 0.152, Negative binomial regression model; Model included the randomised treatment group as the independent variable and duration of time in study as an offset; Incidence rate ratio = 1.48, 95% CI 2-sided [0.86 to 2.53], Standard Error of Mean 0.40 — A rate ratio <1 favours SZC compared to SoC

5. Secondary Outcome: Time to First Occurrence of RAASi Down-titration (or Discontinuation) at Any Time Post-discharge up to 180 Days
Description: The time to first occurrence of RAASi down-titration (or discontinuation) was calculated as date of first occurrence of (RAASi down-titration, all-cause death, date of loss to follow-up) - date of randomization + 1.
  The median time to event (days) is presented.
Time Frame: At any time post-discharge (from Visits 4 to 10), up to 180 days
Population: FAS. The FAS included all randomised participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A: SZC | Arm B: SoC
Number analyzed (Participants) | 68 | 69
Days | NA [NA to NA] — Fewer than 50% of participants experienced an event and no median time, lower confidence interval, and upper confidence interval could be calculated. | NA [NA to NA] — Fewer than 50% of participants experienced an event and no median time, lower confidence interval, and upper confidence interval could be calculated.
Statistical Analysis 1: Comparison: Arm A: SZC vs Arm B: SoC; Test type: Equivalence — This outcome is unpowered; p = 0.515, Regression, Cox; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.50 to 4.35] — An HR <1 favoured SZC to be associated with a longer time to first component of composite endpoint than SoC

6. Secondary Outcome: Time to First Occurrence of Hospital Admission or ED Visit, Both With HK as a Contributing Factor at Any Time Post-discharge up to 180 Days
Description: The time to first occurrence of hospital admission or ED visit, both with HK as a contributing factor, was calculated as date of first occurrence of (Hospital admission or ED visit with HK as a contributing factor, all-cause death, use of rescue therapy for HK, date of loss to follow-up) - date of randomization + 1.
  The median time to event (days) is presented.
Time Frame: At any time post-discharge (from Visits 4 to 10), up to 180 days
Population: FAS. The FAS included all randomised participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A: SZC | Arm B: SoC
Number analyzed (Participants) | 68 | 69
Days | NA [NA to NA] — Fewer than 50% of participants experienced an event and no median time, lower confidence interval, and upper confidence interval could be calculated. | NA [NA to NA] — Fewer than 50% of participants experienced an event and no median time, lower confidence interval, and upper confidence interval could be calculated.
Statistical Analysis 1: Comparison: Arm A: SZC vs Arm B: SoC; Test type: Equivalence — This outcome is unpowered; p = 0.258, Regression, Cox; [statistical method as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.07 to 1.83] — An HR <1 favoured SZC to be associated with a longer time to first component of composite endpoint than SoC

7. Secondary Outcome: Number of Events (Hospital Admissions or ED Visits) With HK as a Contributing Factor, at Any Time Post-discharge up to 180 Days
Description: The number of events (hospital admissions or ED visits) with HK as a contributing factor, at any time post-discharge up to 180 days is presented.
  Participants who discontinued treatment, used rescue therapy for HK, experienced all-cause death or loss to follow-up prior to 180 days post-discharge or who downtitrated (including discontinued) RAASi were to have all available hospital admission data used irrespective of the intercurrent event (treatment policy strategy).
Time Frame: At any time post-discharge (from Visits 4 to 10), up to 180 days
Population: FAS. The FAS included all randomised participants.
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Arm A: SZC | Arm B: SoC
Number analyzed (Participants) | 68 | 69
Events | 0.1 (0.24) | 0.1 (0.26)
Statistical Analysis 1: Comparison: Arm A: SZC vs Arm B: SoC; Test type: Equivalence — This outcome is unpowered; p = 0.239, Negative binomial regression model; Model included the randomised treatment group as the independent variable and duration of time in study as an offset; Incidence risk ratio = 0.42, 95% CI 2-sided [0.10 to 1.81], Standard Error of Mean 0.31 — A rate ratio <1 favours SZC compared to SoC

ADVERSE EVENTS:
Time Frame: Inpatient period (IP): included treatment-emergent adverse events (TEAEs; including serious adverse events [SAEs]) during the IP up to randomization. and adverse events (AEs) prior to first dose that worsened post-dose, up to 14 days Outpatient period (OP): Included TEAEs (including SAEs) during the OP up to 7 days after last dose, and AEs prior to first dose that worsened post-dose, up to approximately 6 months
Description: The AEs that occurred during the IP and OP are reported.
  IP: Safety Set Open. Of the 186 participants enrolled, 12 participants did not receive 1 dose of SZC during the IP and were excluded from the analysis.
  OP: Safety Set Randomized. Of the 137 participants randomized (68 to Arm A and 69 to Arm B), there was 1 participant in Arm B who did not receive treatment during the OP and was excluded from the analysis.
Groups:
- Inpatient Period: Participants were treated with SZC as per local label (correction and/or maintenance treatment), starting at baseline and based on local K+ measurement obtained within 24 hours of treatment initiation.
Arm/Group | Inpatient Period | Outpatient Period - Arm A: SZC | Outpatient Period - Arm B: SoC
All-Cause Mortality (participants affected / at risk) | 2/174 | 6/68 | 2/68
Serious Adverse Events (participants affected / at risk) | 10/174 | 29/68 | 21/68
Other Adverse Events (participants affected / at risk) | 0/174 | 22/68 | 30/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatient Period (N=174) | Outpatient Period - Arm A: SZC (N=68) | Outpatient Period - Arm B: SoC (N=68)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 1 (2)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Penile abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (4) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myasthenia gravis crisis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (5) | 2 (3)
Male genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inpatient Period (N=174) | Outpatient Period - Arm A: SZC (N=68) | Outpatient Period - Arm B: SoC (N=68)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 8 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 6 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 12 (14) | 17 (19)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 4 (4)
Renal impairment (Renal and urinary disorders) | 0 (0) | 5 (5) | 4 (4)
Cardiac failure (Cardiac disorders) | 0 (0) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
Results should be interpreted with great caution due to a high and imbalanced missingness of K+ results from the central laboratory at Day 180 / Visit 10 (51.5% in the SZC group and 36.2% in the SoC group). Hence, results are only described with no conclusive statement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT05347693/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT05347693/SAP_001.pdf